CLINICAL TRIAL: NCT00199901
Title: Randomized, Double-blind Phase II Trial of NY-ESO-1 ISCOMATRIX® Vaccine and ISCOMATRIX® Adjuvant Alone in Patients With Resected Stage Ilc, Illb, lIIc, or IV Malignant Melanoma
Brief Title: Study of NY-ESO-1 ISCOMATRIX® in Patients With High-risk, Resected Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUD2003-009
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Melanoma
Keywords: Phase II; Randomized Controlled Trial; Double-Blind; Cancer Vaccine; NY-ESO-1 protein, human; ISCOMATRIX®, immunological adjuvant
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Active Comparator): NY-ESO-1 ISCOMATRIX® vaccine
  Interventions: Biological: NY-ESO-1 ISCOMATRIX®
- Adjuvant Alone (Placebo Comparator): ISCOMATRIX® adjuvant alone
  Interventions: Biological: ISCOMATRIX® adjuvant

INTERVENTIONS:
Biological: NY-ESO-1 ISCOMATRIX® — 100 μg of NY-ESO-1 protein formulated with 120 μg of ISCOMATRIX® adjuvant.
  Each patient will receive four intramuscular injections of NY-ESO-1 ISCOMATRIX® vaccine. The first three doses will be given at four-week intervals, days 1, 29, and 57, (± 3 days of scheduled date). The fourth injection will be given at month 6 (day 183 ± 3 days).
  Arms: Vaccine
Biological: ISCOMATRIX® adjuvant — 120 μg of ISCOMATRIX® adjuvant
  Each patient will receive four intramuscular injections of ISCOMATRIX® adjuvant alone. The first three doses will be given at four-week intervals, days 1, 29, and 57, (± 3 days of scheduled date). The fourth injection will be given at month 6 (day 183 ± 3 days).
  Arms: Adjuvant Alone

SUMMARY:
The purpose of this trial is to assess whether treatment with NY-ESO-1 ISCOMATRIX® vaccine improves outcomes for people with Malignant Melanoma which has been removed, but is at high risk of relapse.

DETAILED DESCRIPTION:
NY-ESO-1 protein is an immune target found in many cancers including melanoma. ISCOMATRIX® adjuvant enhances immune responses. This trial compares NY-ESO-1 ISCOMATRIX® vaccine with ISCOMATRIX® adjuvant alone to assess whether treatment with NY-ESO-1 ISCOMATRIX® vaccine improves outcomes for participants with Malignant Melanoma which has been removed, but is at high risk of recurrence.

Eligible participants are randomly allocated to a treatment arm. Treatment involves four intramuscular (into a muscle) injections (1 injection every 4 weeks x 3, plus 1 injection at 6 months).

Participants are assessed for recurrence of melanoma, safety and immune responses (by blood test) over the 18 month study period. Off study, their own doctor will follow them for melanoma recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignant melanoma.
* Tumor expression of NY-ESO-1 antigen by immunohistochemistry.
* Fully resected AJCC stage IIc, IIIb, IIIc or IV melanoma.
* Within six months of surgery for melanoma.
* Full recovery from surgery.
* No immunotherapy or systemic adjuvant therapy for melanoma since most recent relapse and/or resection. (Previous adjuvant therapy accepted providing patient relapsed and resected after this.)
* Age 18 years or older.
* Able to give written informed consent.
* Vital laboratory parameters within normal range, or protocol specified ranges.

Exclusion Criteria:

* Other serious or significant illnesses.
* Resected cerebral metastases.
* Ocular melanoma.
* Other malignancy within last 3 years, except for treated non-melanoma skin cancer and cervical cancer in situ.
* Using immunosuppressive drugs.
* Anticoagulation.
* Known HIV positivity.
* Chemotherapy or radiation therapy in last four weeks (6 weeks for nitrosourea drugs).
* Not available for immunological and clinical follow-up assessments.
* Participation in prior clinical trial involving an investigational agent within last 4 weeks.
* Previous isolated limb perfusion (ILP).
* Pregnancy or breastfeeding.
* Refusal or inability to use effective means of contraception for women of childbearing potential.
* Mental impairment that may compromise ability to give informed consent and to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jonathan S Cebon, MBBS PhD, Study Chair — Ludwig Institute for Cancer Research; Prof. Martin Gore, MBBS PhD, Principal Investigator — The Royal Marsden Hospital
Locations (15):
- Australia (6):
  - Sydney Melanoma Unit - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Newcastle Melanoma Unit - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Mater Medical Centre, Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Health (Ludwig Institute Oncology Unit), Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- University of Auckland (Waitemata DHB), Auckland, New Zealand
- United Kingdom (8):
  - University Hospital - Birmingham, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Western Infirmary, Glasgow
  - St Georges Hospital, London
  - Royal Marsden Hospital, London
  - Mount Vernon Hospital, Northwood
  - Weston Park Hospital, Sheffield
  - Southampton University Hospitals, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with resected Stage IIc, lIIb, IIIc and IV melanoma who met eligibility requirements were randomized and stratified by stage of disease to receive 4 intramuscular injections of either NY-ESO-1 ISCOMATRIX® or ISCOMATRIX® adjuvant.
  The first patient was dosed on 27Sep2005 and the last dose was on 27Jun2007.
Pre-assignment Details: 111 patients were screened and randomized. One patient did not receive study drug. 56 patients were randomized to the NY-ESO-1 ISCOMATRIX® arm and 54 to the ISCOMATRIX® adjuvant arm.
Groups:
- NY-ESO-1 ISCOMATRIX® Vaccine: 100 μg of NY-ESO-1 protein formulated with 120 μg of ISCOMATRIX® adjuvant. Each patient received four intramuscular injections of NY-ESO-1 ISCOMATRIX® vaccine. The first three doses were given at four-week intervals, days 1, 29, and 57, (± 3 days of scheduled date). The fourth injection was given at month 6 (day 183 ± 3 days).
- ISCOMATRIX® Adjuvant: 120 μg of ISCOMATRIX® adjuvant. Each patient received four intramuscular injections of ISCOMATRIX® adjuvant. The first three doses were given at four-week intervals, days 1, 29, and 57, (± 3 days of scheduled date). The fourth injection was given at month 6 (day 183 ± 3 days).
Period: Overall Study
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Started | 56 | 54
Completed | 29 | 30
Not Completed | 27 | 24
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Progressive Disease | 24 | 24

BASELINE CHARACTERISTICS:
Population: All patients randomized and received NY-ESO-1 ISCOMATRIX® Vaccine or ISCOMATRIX® adjuvant.
Groups:
- Total: Total of all reporting groups
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.28) | 53.0 (13.90) | 53.7 (13.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 37 | 32 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 54 | 51 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 56 | 54 | 110
Region of Enrollment [Number; unit: participants]
  New Zealand | 2 | 4 | 6
  United Kingdom | 17 | 15 | 32
  Australia | 37 | 35 | 72
ECOG [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    ECOG PS 0 | 51 | 44 | 95
    ECOG PS 1 | 2 | 8 | 10
    ECOG PS 2 | 0 | 0 | 0
    ECOG PS 3 | 0 | 0 | 0
    ECOG PS 4 | 0 | 0 | 0
    Not Recorded | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate of Relapse-free Survival at 18 Months
Description: The number of patients who were alive and relapse free 18 months after starting therapy and the number of patients who relapsed or died within 18 months of starting therapy.
  Disease was assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) as measured by CT. Disease progression or relapse was based on an increase of 20% or more in the sum of the longest diameter of target lesions, the appearance of any new lesion as confirmed by CT scan or death.
Time Frame: 18 months
Population: All randomized patients who received at least one dose of NY-ESO-1 ISCOMATRIX® vaccine or ISCOMATRIX® adjuvant.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 56 | 54
Participants
  Number of patients relapse free at 18 months | 29 | 28
  Number of patients relapsed at 18 months | 27 | 26
Statistical Analysis 1: Comparison: NY-ESO-1 ISCOMATRIX® Vaccine vs ISCOMATRIX® Adjuvant; Test type: Superiority; Hazard Ratio (HR) = 0.913, 95% CI 2-sided [0.532 to 1.568]

2. Secondary Outcome: Number of Patients With Treatment -Emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Adverse events (AEs) were reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, electrocardiograms, magnetic resonance imaging, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 18 months. AEs were considered to be treatment emergent (TEAE) if they occurred or worsened in severity after the first dose of study treatment.
Time Frame: 18 months
Population: All randomized patients who received at least one dose of NY-ESO-1 ISCOMATRIX® vaccine or ISCOMATRIX® adjuvant.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 56 | 54
Participants
  Number of subjects with at least one TEAE | 54 | 52
  Number of subjects with SAE | 10 | 12
  Number of subjects discontinued due to TEAE | 2 | 7

3. Secondary Outcome: Relapse-Free Survival During the Entire Period of Observation (up to 6 Years).
Description: Disease was assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) as measured by CT. Disease progression or relapse was based on an increase of 20% or more in the sum of the longest diameter of target lesions, the appearance of any new lesion as confirmed by CT scan or death.
Time Frame: through study completion; up to 6 years
Population: All patients who received at least one dose of NY-ESO-1 ISCOMATRIX® vaccine or ISCOMATRIX® adjuvant.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 56 | 54
Participants
  Number of Patients who did not relapse | 23 | 25
  Number of patients who relapsed | 33 | 29
Statistical Analysis 1: Comparison: NY-ESO-1 ISCOMATRIX® Vaccine vs ISCOMATRIX® Adjuvant; Test type: Superiority; Hazard Ratio (HR) = 0.880, 95% CI 2-sided [0.532 to 1.455]

4. Secondary Outcome: Overall Survival
Description: Overall Survival measured during the entire Period of Observation (up to 6years).
  Overall survival was measured from start of treatment to the last follow-up or death.
Time Frame: through study completion; up to 6 years
Population: All randomized patients who received at least one dose of NY-ESO-1 ISCOMATRIX® vaccine or ISCOMATRIX® adjuvant.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 56 | 54
Participants
  Number of Patients Alive at last follow-up | 32 | 31
  Number of Patients Dead at last follow-up | 24 | 23
Statistical Analysis 1: Comparison: NY-ESO-1 ISCOMATRIX® Vaccine vs ISCOMATRIX® Adjuvant; Test type: Superiority; Hazard Ratio (HR) = 0.911, 95% CI 2-sided [0.514 to 1.614]

5. Secondary Outcome: NY-ESO-1 Antibody Response at Baseline Reported on a Scale of 0 to 4 With 0 Being no or Minimal Antibody Response and 4 the Highest Antibody Response
Description: NY-ESO-1-specific antibodies were measured by an enzyme-linked immunosorbent assay ( ELISA) method at baseline and on days 71, 197, 365 and end of study. The results are reported as antibodies to NY-ESO-1-specific Total IgG (reciprocal titer) and were scored on a scale of 0-4 with 0 being no or minimal antibody response (reciprocal titer of 0-100) and 4 a strong antibody response (reciprocal titer of >100,000). The number of patients with each antibody response level are tabulated at each timepoint.
Time Frame: Baseline
Population: All randomized patients who received at least one dose of NY-ESO-1 ISCOMATRIX® vaccine or ISCOMATRIX® adjuvant and provided blood samples for analysis at the required time. Patients who discontinued the study prior to the scheduled day were not included at the later timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 46 | 45
Participants
  0 | 31 | 32
  1 | 2 | 0
  2 | 8 | 10
  3 | 3 | 2
  4 | 2 | 1

6. Secondary Outcome: NY-ESO-1 Antibody Response on Day 71 Reported on a Scale of 0 to 4 With 0 Being no or Minimal Antibody Response and 4 the Highest Antibody Response
Description: as for outcome 5
Time Frame: Day 71
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 43 | 45
Participants
  0 | 0 | 32
  1 | 0 | 2
  2 | 2 | 8
  3 | 32 | 2
  4 | 9 | 1

7. Secondary Outcome: NY-ESO-1 Antibody Response on Day 197 Reported on a Scale of 0 to 4 With 0 Being no or Minimal Antibody Response and 4 the Highest Antibody Response
Description: as for outcome 5
Time Frame: Day 197
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 34 | 32
Participants
  0 | 0 | 20
  1 | 0 | 0
  2 | 3 | 7
  3 | 21 | 5
  4 | 10 | 0

8. Secondary Outcome: NY-ESO-1 Antibody Response on Day 365 Reported on a Scale of 0 to 4 With 0 Being no or Minimal Antibody Response and 4 the Highest Antibody Response
Description: as for outcome 5
Time Frame: Day 365
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 27 | 29
Participants
  0 | 0 | 19
  1 | 1 | 0
  2 | 3 | 6
  3 | 22 | 4
  4 | 1 | 0

9. Secondary Outcome: NY-ESO-1 Antibody Response at End of Study Reported on a Scale of 0 to 4 With 0 Being no or Minimal Antibody Response and 4 the Highest Antibody Response
Description: as for outcome 5
Time Frame: End of Study (month 18)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
Number analyzed (Participants) | 37 | 36
Participants
  0 | 0 | 26
  1 | 2 | 2
  2 | 6 | 4
  3 | 26 | 4
  4 | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were documented from informed consent through 18 months (regardless of causality to study drug).
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Adverse events (AEs) were documented from the time informed consent was signed through 18 months. AEs were considered to be treatment emergent (TEAE) if they occurred or worsened in severity after the first dose of study treatment.
Arm/Group | NY-ESO-1 ISCOMATRIX® Vaccine | ISCOMATRIX® Adjuvant
All-Cause Mortality (participants affected / at risk) | 24/56 | 23/54
Serious Adverse Events (participants affected / at risk) | 10/56 | 12/54
Other Adverse Events (participants affected / at risk) | 54/56 | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO-1 ISCOMATRIX® Vaccine (N=56) | ISCOMATRIX® Adjuvant (N=54)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Abdominal neoplasm (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 1
Malignant melanoma (Skin and subcutaneous tissue disorders) | 2 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Mass excision (Surgical and medical procedures) | 3 | 2
Radioactive iodine therapy (Surgical and medical procedures) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 1 | 0
Cerebral artery stenosis (Vascular disorders) | 0 | 1
Transient ischemic attack (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO-1 ISCOMATRIX® Vaccine (N=56) | ISCOMATRIX® Adjuvant (N=54)
lymphadenopathy (Blood and lymphatic system disorders) | 4 | 1
nausea (Gastrointestinal disorders) | 9 | 7
chills (General disorders) | 6 | 1
fatigue (General disorders) | 13 | 16
influenza like illness (General disorders) | 26 | 9
injection site discomfort (General disorders) | 5 | 1
injection site erythema (General disorders) | 9 | 1
injection site pain (General disorders) | 28 | 17
injection site reaction (General disorders) | 16 | 11
lethargy (General disorders) | 5 | 3
malaise (General disorders) | 3 | 0
pyrexia (General disorders) | 6 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6
back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 6
headache (Nervous system disorders) | 18 | 13
cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4
rash (Skin and subcutaneous tissue disorders) | 4 | 5
mass excision (Surgical and medical procedures) | 3 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 5
diarrhea (Gastrointestinal disorders) | 1 | 3
mass (General disorders) | 1 | 3
influenza (Respiratory, thoracic and mediastinal disorders) | 1 | 3
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 3
dizziness (Nervous system disorders) | 2 | 3
paresthesia (Nervous system disorders) | 1 | 3
skin lesion excision (Surgical and medical procedures) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No